CLINICAL TRIAL: NCT00524524
Title: An Exploratory Biomarker Study of ARQ 501 in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ArQule, Inc., a subsidiary of Merck Sharp & Dohme LLC, a subsidiary of Merck & Co., Inc. (Rahway, NJ USA) (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARQ 501-109
Record Dates: First submitted 2007-08-30; First posted 2007-09-03 (Estimated); Last update posted 2011-10-19 (Estimated); Status verified 2011-10

CONDITIONS: Advanced Solid Tumors
Keywords: solid tumors; biopsy
MeSH Terms: interventions — beta-lapachone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ARQ 501 — Weekly IV Infusion; 450 mg/m2

SUMMARY:
This study is designed to evaluate the response of several biomarkers in patients treated with ARQ 501. The results of the study may help the sponsor understand the effect of the study drug on these biomarkers and their respective role in cancer growth control.

DETAILED DESCRIPTION:
ARQ 501 is an investigational anticancer agent that consists of a fully synthetic small molecule version of β-lapachone (3,4-dihydro-2,2-dimethyl-2H-naphtho[1,2-b]pyran-5,6-dione) in a stable formulation for intravenous (IV) administration. ARQ 501 selectively induces apoptosis in cancer cells by the direct activation of the cellular checkpoints without damaging deoxyribonucleic acid (DNA) or microtubules. This therapeutic approach is known as Activated Checkpoint Therapy (ACT)sm. ACTsm is a novel strategy for treating and preventing cancers. Cell cycle checkpoints constitute an internal surveillance system that detects cellular, especially genetic, damage and either allows the cells to repair the damage, or induces apoptosis when damage is not repairable. Cancer cells are selectively eliminated upon checkpoint activation due to presence of irreparable DNA damage. It is believed that the rapid and selective induction of apoptosis in cancer cells by ARQ 501 is caused by a correspondingly rapid and sustained increase of the pro-apoptotic protein E2F1.

Preclinical studies have shown that exposure to ARQ 501 results in the activation or inactivation of a panel of 5 biomarkers. Time course changes in human tumor xenograft biomakers in athymic mice after exposure to ARQ 501 can be classified into 3 biomarker groups: those that changed shortly after exposure and returned to normal within 24 hours; those that changed shortly after exposure and remained for 24 hours or longer; and those that changed after 24 hours or later.

The primary objective is to evaluate the response of biomarkers in patients treated with ARQ 501. The exploratory study will help to illuminate the pharmacodynamics of these biomarkers, their roles in the cancer growth control, and their potential predictive or prognostic values for the disease and treatment of ARQ 501 in humans.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide signed and dated informed consent prior to study-specific screening procedures.
2. Patients must have histologically or cytologically confirmed advanced solid tumor(s).
3. Measurable disease as defined by RECIST (see Section 9.0).
4. Patients must have Karnofsky performance status (KPS) ≥ 70%.
5. Male or female patients of child-producing potential must agree to contraception or avoidance of pregnancy measures during the study and for 30 days after the infusion of ARQ 501.
6. Females of childbearing potential must have a negative serum pregnancy test within seven days prior to the administration of study drug.
7. ≥ 18 years old.
8. Hemoglobin ≥ 10 g/dL
9. Absolute neutrophil count (ANC) ≥ 1.5 x 10 9/L (≥1,500/mm3).
10. Platelets ≥ 100 x 10 9/L (≥ 100,000/mm3).
11. Total bilirubin ≤ 1.5 x upper limit of normal (ULN) or ≤ 3.0 x ULN with metastatic liver disease.
12. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN or ≤ 5.0 x ULN with metastatic liver disease.
13. Creatinine ≤ 1.5 × ULN

Exclusion Criteria:

1. Active, uncontrolled systemic infection considered opportunistic, life threatening or clinically significant at the time of treatment
2. Received anticancer chemotherapy, immunotherapy, radiotherapy, surgery or investigational agents within four weeks of first infusion
3. Symptomatic or untreated central nervous system (CNS) involvement
4. Previous exposure to ARQ 501

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2007-08; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the pharmacodynamics of a panel of biomarkers following administration of ARQ 501 | Up to 30 hours after a single dose of ARQ 501

SECONDARY OUTCOMES:
To further characterize the safety and tolerability of ARQ 501
To assess anti-tumor activity of ARQ 501

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Shapiro, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States